CLINICAL TRIAL: NCT05307302
Title: The Relationship Between Elbow Proprioception, Upper Extremity Physical Performance, and Passing Accuracy in Adolescent Basketball Players
Brief Title: Proprioception, Physical Performance, and Passing Accuracy in Adolescent Basketball Players
Status: Completed | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Hakan AKKAN, PhD, PT, Kutahya Health Sciences University
Other Study IDs: KutahyaHSU-002
Record Dates: First submitted 2022-03-24; First posted 2022-04-01 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Basketball Players
Keywords: proprioception; elbow; physical performance; passing accuracy; adolescent

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adolescent basketball players: Adolescent basketball players between the ages of 13-18 playing in basketball teams
  Interventions: Diagnostic Test: Force Sense; Diagnostic Test: Joint Reproduction Sense; Diagnostic Test: Seated Medicine Ball Throw; Diagnostic Test: Closed Kinetic Chain Upper Extremity Stability Test; Diagnostic Test: Passing Accuracy

INTERVENTIONS:
Diagnostic Test: Force Sense — A measure of proprioception, using a handheld dynamometer (MicroFET2-hoggan Health Industries Inc.), in a sitting position in a standardized position of the elbow joint of the dominant upper extremity (90 degree of flexion). Measurement of the elbow joint flexion force sense will be expressed as percentages. Each of the targeted trials will be calculated as a percentage of the maximum voluntary contraction (MVC) reference measure. The difference between the targeted and the actual percentage of MVC for each of the trials will be then calculated as a percentage of the targeted MVC, to reflect the proportion of error.
Diagnostic Test: Joint Reproduction Sense — A measure of proprioception, using a smart phone goniometer (Android Clinometer) application, in a sitting position in a standardized position of the elbow joint of the dominant upper extremity. Measurement of the elbow joint position reproduction will be expressed as degrees of reproduced angle. Absolute Error (AE) score will be calculated by the absolute value of the difference in degrees of the angle reproduced after subtracting the angle targeted.
Diagnostic Test: Seated Medicine Ball Throw — A measure of upper limb physical performance, using 2-kg medicine ball and a standardized protocol, throwing distance expressed in meters.
Diagnostic Test: Closed Kinetic Chain Upper Extremity Stability Test — A measure of upper limb physical performance, using body weight and a standardized protocol, touches between hands expressed in number of touches.
Diagnostic Test: Passing Accuracy — A measure of the basketball passing skills, passing of The American Alliance for Health, Physical Education, Recreation and Dance (AAHPERD) test battery will be used in a standardized protocol. Accurate passes will be expressed in points.

SUMMARY:
The relationship between elbow proprioception, upper extremity physical performance, and passing accuracy in adolescent basketball players will be explored.

DETAILED DESCRIPTION:
Proprioception is defined as transmitting the sense of the position of our body, interpreting incoming information about posture, and performing the movement to be done consciously or unconsciously. It is critical in controlling and coordinating goal-directed multi-joint movements. It is crucial to learn and perform the sport-specific techniques correctly to increase performance in training and competitions.

Recently, the interest in basketball has increased, and the number of adolescents participating in this sport has increased at the same rate. Passing is the most widely used technical skill after shooting in basketball. A basketball player's performance and a team's success mainly depend on their passing skills. Because passing in basketball is one of the important actions in the game. It has been stated that the error/success ratio of the player on the passing skill is the main distinguishing factor between beginners and experienced players in competitions.

For this reason, the performance and season-long success of the players in basketball depend mainly on their passing skills. The Physical Performance Tests can be used to determine functional performance and evaluate progression in athletic populations. It has become necessary to conduct studies investigating basketball passing to improve training capacity, the performance, and skills of players.

Some studies in the literature investigate the possible relationship between proprioception and sportive success. One of them emphasized the relationship between free throw percentage and shoulder joint position sense. They also stated that proprioceptive exercises (especially above 90° of the shoulder ROM) could be included in the training program to increase the percentage of free throws. On the other hand, one study examined the relationship between basketball players' free-throw performance, elbow, and wrist joint position sense and found a moderate correlation between free-throw success rate and wrist and elbow joint position sense.

The studies on upper extremity proprioception in basketball players mainly focus on examining free-throw performance, and there is no study examining the relationship between proprioception and passing accuracy. In addition, no research has been found exploring the relationship between upper extremity physical performance and proprioception in basketball. Therefore, this study hypothesizes that a player with good elbow proprioception and upper extremity physical performance tests would have high pass accuracy, considering the importance of passing in basketball.

ELIGIBILITY:
Inclusion Criteria:

* Those who are between the ages of 13-18
* Those who have licensed active basketball players
* Having verbal and written communication skills in Turkish

Exclusion Criteria:

* Refusal
* Having had any upper extremity surgery
* Having a diagnosis of any upper extremity musculoskeletal conditions

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adolescent basketball players in amateur basketball club teams in Kütahya Province will be recruited for this study.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2022-08-16 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Force Sense | At baseline
  A measure of proprioception, using a handheld dynamometer, in a sitting position in a standardized position of the elbow joint of the dominant upper extremity (90 degree of flexion).
Joint Position Reproduction | At baseline
  A measure of proprioception, using a smart phone goniometer (Android Clinometer) application, in a sitting position in a standardized position of the elbow joint of the dominant upper extremity.
Seated Medicine Ball Throw | At baseline
  A measure of upper limb physical performance, using body weight and a standardized protocol, touches between hands expressed in number of touches.
Closed Kinetic Chain Upper Extremity Stability Test | At baseline
  A measure of upper limb physical performance, using body weight and a standardized protocol, touches between hands expressed in number of touches.
Passing Accuracy | At baseline
  A measure of the basketball passing skills, passing of The American Alliance for Health, Physical Education, Recreation and Dance (AAHPERD) test battery will be used in a standardized protocol. Accurate passes will be expressed in points.

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Akkan, PT, PhD, Principal Investigator — Kutahya Health Sciences University
Locations (1):
- Kutahya Health Sciences University, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Proske U. Exercise, fatigue and proprioception: a retrospective. Exp Brain Res. 2019 Oct;237(10):2447-2459. doi: 10.1007/s00221-019-05634-8. Epub 2019 Aug 30. PMID 31471677
- [Background] Wright ML, Adamo DE, Brown SH. Age-related declines in the detection of passive wrist movement. Neurosci Lett. 2011 Aug 15;500(2):108-12. doi: 10.1016/j.neulet.2011.06.015. Epub 2011 Jun 17. PMID 21704124
- [Background] Maimon AQ, Courel-Ibanez J, Ruiz FJR. The Basketball Pass: A Systematic Review. J Hum Kinet. 2020 Jan 31;71:275-284. doi: 10.2478/hukin-2019-0088. eCollection 2020 Jan. PMID 32148591
- [Background] Sevrez V, Bourdin C. On the Role of Proprioception in Making Free Throws in Basketball. Res Q Exerc Sport. 2015;86(3):274-80. doi: 10.1080/02701367.2015.1012578. Epub 2015 Mar 16. PMID 25775217
- [Background] Gomez MA, Lorenzo A, Ortega E, Sampaio J, Ibanez SJ. Game Related Statistics Discriminating Between Starters and Nonstarters Players in Women'S National Basketball Association League (WNBA). J Sports Sci Med. 2009 Jun 1;8(2):278-83. eCollection 2009. PMID 24149538